CLINICAL TRIAL: NCT01455389
Title: Phase I/II Clinical Trial Combining TUSC2-nanoparticles and Erlotinib in Stage IV Lung Cancer
Brief Title: TUSC2-nanoparticles and Erlotinib in Stage IV Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Trial terminated by sponsor after decision to evaluate combination of quaratusugene ozeplasmid and osimertinib instead of further evaluating quaratusugene ozeplasmid and erlotinib.
Sponsor: Genprex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-002
Record Dates: First submitted 2011-10-17; First posted 2011-10-20 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Non-small cell lung cancer; NSCLC; FUS1-nanoparticles; DOTAP:Chol-TUSC2; DOTAP:Cholesterol-TUSC2 Liposome Complex; Erlotinib; Erlotinib Hydrochloride; OSI-774; Tarceva; Dexamethasone; Decadron; Diphenhydramine; Benadryl; Benylin Cough SyrupPharmacokinetic; PK
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Dexamethasone; Calcium Dobesilate; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DOTAP + Erlotinib (Experimental): DOTAP:Chol-TUSC2 0.045 mg/kg by vein over 25-35 minutes on day 1 of each 21 day cycle; and Erlotinib 100 mg by mouth daily for each 21 day cycle.
  Interventions: Drug: DOTAP:Chol-TUSC2; Drug: Erlotinib; Drug: Dexamethasone; Drug: Diphenhydramine

INTERVENTIONS:
Drug: DOTAP:Chol-TUSC2 — Starting Dose 0.045 mg/kg by vein on day 1 of each 21 day cycle; Phase II is Maximum Tolerated Dose from Phase I.
  Other Names: DOTAP:Cholesterol-TUSC2 Liposome Complex
Drug: Erlotinib — Starting Dose 100 mg by mouth each day of a 21 day cycle (except for first week of Cycle 1, if enrolled in Phase II delayed-schedule group). Phase II is Maximum Tolerated Dose from Phase I.
  Other Names: Erlotinib Hydrochloride; OSI-774; Tarceva
Drug: Dexamethasone — 8 mg orally 24 and 12 hours and 20 mg by vein 30 minutes before DOTAP:Chol-TUSC2 treatment followed by 8 mg orally at 12, 24 and 36 hours after treatment (total number doses = 5).
  Other Names: Decadron
Drug: Diphenhydramine — 50 mg by mouth or by vein 30 minutes prior to treatment with DOTAP:Chol TUSC2
  Other Names: Benadryl; Benylin Cough Syrup [OTC]

SUMMARY:
The goal of phase 1 of this clinical research study is to find the highest dose of DOTAP:Chol-TUSC2 that can be safely given in combination with Tarceva (erlotinib hydrochloride) to patients with NSCLC.

The goal of phase 2 of this clinical research study is to learn if the combination of DOTAP:Chol-TUSC2 and erlotinib hydrochloride can help to control NSCLC.

The safety of this drug combination will also be studied in both phases.

DOTAP:Chol-TUSC2 (previously FUS1) is a drug that helps transfer a gene called TUSC2 into cancer cells. Researchers think that cells without this gene may be involved in the development of lung cancer tumors. They want to find out if replacing the gene in these cells may keep the tissue from forming cancer cells.

Erlotinib hydrochloride is designed to block a protein on tumor cells that may control tumor growth and survival. This may stop tumors from growing.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of DOTAP:Chol-TUSC2 and erlotinib hydrochloride based on when you join this study. Up to 4 dose levels of the study drug combination will be tested. Three (3) participants will be enrolled at each dose level. The first group of participants will receive the first dose combination level. After this dose is given, the participants will be watched for 3 weeks to check for any serious side effects at that dose level. If any participants in this first group have intolerable side effects, 1-2 lower dose combinations of the study drugs may be tested.

If no intolerable side effects are seen in the first group, the second study group will receive the next planned dose combination. If no intolerable side effects are seen in this group, the last dose combination will be tested.

If you are enrolled in the Phase II portion, you will receive the highest study combination dose that was tolerated in the Phase I portion.

During the Phase II portion of the study, half of the participants will not start receiving erlotinib hydrochloride until Day 8 of Cycle 1 (+/- 1 day). Every odd-numbered participant (1, 3, 5, and so on) enrolled in Phase II will receive this delayed schedule for erlotinib hydrochloride. NOTE: For all participants dosing of erlotinib has been changed to begin on Day 8 of Cycle 1 and then daily.

Study Drug Administration:

You will receive the drugs dexamethasone and diphenhydramine before each infusion of DOTAP:Chol-TUSC2, to try to lower the risk of possible allergic reactions to the study drug. Dexamethasone will be given by mouth about 24 hours before your dose of DOTAP:Chol-TUSC2, and by vein about 30 minutes before the dose. Diphenhydramine will also be given (either by mouth or as an injection) about 30 minutes before the dose.

DOTAP:Chol-TUSC2 is given by vein as an infusion over 25-35 minutes, on Day 1 of every 3-week study cycle.

You will take erlotinib hydrochloride by mouth in tablet form every day you are on study (except for first week of Cycle 1, if you were enrolled in the Phase II delayed-schedule group).

Erlotinib hydrochloride tablets should be taken at about the same time each day. Each erlotinib dose should be taken with about 8 ounces of water, and should be taken 1 hour before or 2 hours after meals. The whole dose must be taken at one time. If you vomit after taking the tablet(s), you should only re-take the dose if the tablet(s) can still be seen and counted.

Study Tests:

Each study cycle is 3 weeks.

On Day 1 of each cycle:

* Your vital signs (blood pressure, heart rate, temperature, and breathing rate) will be measured.
* Urine will be collected for routine tests.
* You will have a test to measure the level of oxygen in your blood.

On Day 1 of Cycle 1 only, blood (about 4 tablespoons total) will be drawn before your first dose of DOTAP:Chol-TUSC2 and then about 24 hours later (+/- 4 hours), for research tests to check your immune system.

On Day 2 of each cycle:

* Blood (about 2 teaspoons) will be drawn for routine tests and tests to check your immune system.
* Your vital signs will be recorded, and you will be asked about any side effects you may have.

On Day 7 of Cycle 1, you will have a liquid tumor biopsy for genetic research tests.

On Day 21 of each cycle:

* You will have a physical exam, including measurement of your vital signs.
* Your medical history will be recorded, and you will be asked about any side effects you may be having.
* Blood (about 2 teaspoons) and urine will be collected for routine tests.

On Day 21 of every other cycle (Cycles 2, 4, 6, and so on), you will have either a chest CT or PET/CT scan to check the status of the disease. Other scans may be performed, if your doctor thinks they are needed.

PK Testing:

If you are in Phase 1 and are one of the first 6 participants to be enrolled on this study, blood (about 2 teaspoons each time) will be drawn for pharmacokinetic (PK) testing. PK testing measures the amount of study drug in the body at different time points. PK samples will be drawn during Cycle 1, at the following times:

* Day 1--before the dose of DOTAP:Chol-TUSC2, at 15 and 30 minutes after the dose, and then 1, 3, and 6 hours after the dose
* Day 2
* Day 4
* Day 8
* Day 15

Length of Treatment:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, intolerable side effects occur, or you are unable to follow study directions.

Long-Term Follow-up:

You will be called by the study staff every 3 months after you stop taking the study drugs. The study staff will ask you questions to find out how you are doing and to collect information on any other therapies you have received for cancer. The call should take about 15 minutes.

This is an investigational study. Erlotinib hydrochloride is commercially available and FDA approved for the treatment of non-small-cell lung cancer. At this time, DOTAP:Chol-TUSC2 is only being used in research.

Up to 57 patients will take part in this study. All will be enrolled at MD Anderson as well as additional clinical sites.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented non-small cell lung cancer (NSCLC)
2. Stage IV NSCLC or recurrent NSCLC that is not potentially curable by radiotherapy or surgery. There is no limit to the number or form of prior therapy regimens received, but patients must have received at least one.
3. All subjects must have tumor specimens adequate for analysis of EGFR mutations or have tumor accessible for pretreatment biopsy, and must consent to post-treatment Guardant ctDNA liquid biopsy. Subjects must have specimens adequate for analysis of EGFR mutations (and other clinically relevant biomarkers)
4. All subjects with an activating EGFR mutation (exon 19 deletion or exon 21 L858R mutation) are eligible IF they have progressed following treatment with a first, second, or third generation EGFR inhibitor. All subjects who are EGFR negative or have wild-type EGFR or another non-activating mutation are eligible.
5. ECOG or Zubrod Performance Status ≤1
6. Age ≥18 years
7. Subjects must have voluntarily signed an informed consent in accordance with institutional policies.
8. Female subjects of childbearing potential (non-childbearing is defined as greater than one year post-menopausal or surgically sterilized) must have a Negative serum pregnancy test (serum beta-HCG) ≤7 days of study treatment. Since beta-HCG may be falsely elevated as a result of malignancy, women of child-bearing potential who have an elevated serum beta-HCG level are eligible for enrollment if they have two (2) Transvaginal Ultrasound (TVUS) scans one (1) week apart along with serial beta-HCG levels two (2) weeks apart that are inconsistent with pregnancy and a Gynecology consult to ensure that the beta- HCG level was at a value high enough to see pregnancy with TVUS.
9. Subjects are required to agree to practice effective birth control (i.e., abstinence, intrauterine device for female subjects) during the study period.
10. Subjects must be ≥4 weeks beyond major surgical procedures such as thoracotomy, laparotomy or joint replacement, and must be ≥1.5 weeks beyond minor surgical procedures such as biopsy of subcutaneous tumors, pleuroscopy, etc., and must not have evidence of wound dehiscence, active wound infection, or comparable major residual complications of the surgery. Note: placement of pleurex catheter is not considered minor surgery for this study.
11. ANC >1500/mm3, platelet count >100,000/mm3 ≤14 days of study treatment
12. PT and PTT <1.25 times the institutional upper limit of normal ≤14 days of study treatment
13. Adequate renal function documented by serum creatinine of ≤1.5 mg/dl or calculated creatinine clearance >50 ml/min ≤14 days of study treatment
14. Adequate hepatic function as documented by serum bilirubin <1.5 mg/dl and SGOT and SGPT ≤2.5 X upper limit of normal ≤14 days of study treatment
15. Subjects with asymptomatic brain metastases that have been treated are eligible if the following criteria are met: No history of seizures in the preceding 6 months. Definitive treatment must have been completed ≥4 weeks prior to start of study treatment. Subjects must be off steroids that were being administered because of brain metastases or related symptoms for ≥2 weeks prior to start of study treatment. Post-treatment imaging ≤2 weeks of informed consent must demonstrate stability or regression of the brain metastases.
16. Stable cardiac condition with a left ventricular ejection fraction ≥40% ≤28 days of study treatment

Exclusion Criteria:

1. Subject is female who is pregnant or breast-feeding.
2. Subject received investigational therapy (i.e., agents that are not FDA-approved), including monoclonal antibodies such as bevacizumab or cetuximab, or has received radiotherapy to the skull, spine, thorax or pelvis within ≤30 days of start of study treatment. Subjects are permitted to have received palliative radiotherapy to an extremity provided ≥14 days have elapsed since completion of radiotherapy, provided the subject received ≤10 radiotherapy fractions and a dose ≤30 Gy to that site, and provided skull, spine, thorax or pelvis were not in the radiotherapy field.
3. Subject received standard chemotherapy with FDA-approved agents within ≤21 days of start of study treatment.
4. Subject received a targeted therapy within ≤14 days prior to start of study treatment.
5. Subject has active systemic viral, bacterial or fungal infection(s) requiring treatment.
6. Subject has brain metastases (except as allowed in Section 3.2.1). Neurological assessment will be used to determine brain metastases.
7. Subject has serious concurrent illness or psychological, familial, sociological, geographical, or other concomitant conditions that, in the opinion of the investigator, would not permit adequate follow-up and compliance with the study protocol.
8. Subject received prior gene therapy or cell therapy.
9. Subject has history of myocardial infarction or unstable angina ≤6 months of start of study treatment.
10. Subject is known to be HIV positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-10-27 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) Level for Drug Treatment Combination | First 21 day cycle
  MTD defined as dose level at which less than 2 participants experience dose-limiting toxicity (DLT). Toxicity graded according to National Cancer Institute (NCI) Common Toxicity Criteria (CTC) Version 4. DLT will be grade > 3 toxicity occurring during the first cycle of therapy (i.e., within the first 3 weeks).

SECONDARY OUTCOMES:
Response Rate | After two, 21 day cycles
  Responses determined by RECIST criteria. Responses will include only complete response (CR) + partial response (PR). Participants considered as non-responders when tumor progression by RECIST is observed. Measurable disease is defined as tumor masses with identifiable diameters measurable in two dimensions by computed tomography. Best overall response is best response designation recorded from the start of treatment until disease progression. Complete and partial responses have to be confirmed by two evaluations of the disease taken at least four weeks apart.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Lu, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org